CLINICAL TRIAL: NCT04368273
Title: Phase I Study of Toripalimab Injection (Pd-1 Antibody) With Cisplatin Concurrent IMRT for Local Advanced Cervical Cancer.
Brief Title: Pd-1 Antibody Combined CCRT for Local Advanced Cervical Cancer.
Acronym: CCRT+PD-1
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Junjie Wang, Department director, Peking University Third Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M2019482
Record Dates: First submitted 2020-04-25; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Cervical Cancer
Keywords: PD-1; Radiotherapy; concurrent chemoradiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — spartalizumab; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): PD-1 antibody combined CCRT for patients with local advanced cervical cancer.
  Interventions: Drug: PD-1 antibody

INTERVENTIONS:
Drug: PD-1 antibody — a new treatment drug combined radical radiotherapy concurrent chemotharpy
  Other Names: Toripalimab

SUMMARY:
To evaluate the safety and efficacy of anti-PD-1 (toripalimab) combined with cisplatin concurrent IMRT for locally advanced cervical cancer.

DETAILED DESCRIPTION:
The dose of toripalimab injection (pd-1 antibody) was 240mg/d, d1, i.v. every 14d, totally 4 cycles (56 days)

Concurrent chemoradiotherapy:

Cisplatin 40 mg/m2 i.v., d1, administered once a week; Radiotherapy: pelvic intensity modulated radiotherapy, prescription dose DT: 50.4gy /2Gy/28f;After intraluminal irradiation DT: 30-36 Gy/6Gy/5-6f 2f/w, complete the radiotherapy within 56 days.

Complete at least 4 cycles of concurrent chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. HPV positive in patients with cervical squamous cell carcinoma confirmed by histopathology
2. Patients with local advanced (2018FIGO staged IB3, IIA -IVA) cervical cancer and had not received any treatment before
3. There are measurable lesions according to the efficacy evaluation criteria for solid tumors (RECIST) version 1.1
4. ECOG score 0-2
5. Expected survival ≥3 months
6. LVEF≥55%
7. Bone marrow function: neutrophils ≥1.5×109/L, platelets ≥100×109/L, hemoglobin ≥90g/L
8. Liver and kidney functions: serum creatinine ≤1.5 times the upper limit of normal value;AST and ALT ≤2.5 times normal upper limit or ≤5 times normal upper limit in the presence of liver metastasis;Total bilirubin ≤1.5 times the upper limit of normal value, or ≤2.5 times the upper limit of normal value in patients with Gilbert's syndrome
9. Thyroid function: normal range
10. Non-lactating patients
11. Sign the informed consent

Exclusion Criteria:

1. Patients with previous PD-1 or PD-L1 treatment
2. Patients with previous abdominal or pelvic radiotherapy
3. Other malignant tumors other than cervical cancer appeared in the past 5 years
4. Immunosuppressive drugs were used within 4 weeks prior to the first study treatment, excluding nasal spray, inhaled or other local glucocorticoids or systemic glucocorticoids in physiological doses (i.e., no more than 10 mg/ day prednisone or equivalent doses of other glucocorticoids)
5. Active, known, or suspected autoimmune disease (congenital or acquired)

   ), such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, thyroiditis, etc. (vitiligo or childhood asthma has been completely relieved, adults without any intervention can be included;Patients with type 1 diabetes with good insulin control can also be enrolled, as can hypothyroidism caused by autoimmune thyroiditis that requires hormone replacement therapy.)
6. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation
7. Known allergy to any component of the drug
8. Serious medical diseases that are not under control, such as the combination of serious medical diseases, including severe heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension,uncontrolled infection, active peptic ulcer
9. Received other experimental drugs or participated in other drugs within 30 days of initial administration clinical research on the purpose of anticancer therapy
10. Severe infection occurred within 4 weeks prior to study treatment, including, but not limited to, hospitalization hospital treatment of infection complications, bacteremia or severe pneumonia
11. Human immunodeficiency virus (HIV) positive
12. Hepatitis B surface antigen (HBsAg) positive, and the peripheral blood hepatitis B virus deoxygenation the titer of ribonucleic acid (HBV-DNA) was detected in subjects ≥1×10<3> IU/mL
13. Hepatitis C virus (HCV) antibody positive or human immunodeficiency virus (HIV) Antibody positive and HCV RNA positive

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-05-08 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of acute adverse events | up to 3 months complete treatment
  safety evaluation

SECONDARY OUTCOMES:
Objective response rate | 3 months later after treatment
  efficacy evaluation
Progression-free survival | up to 2 years
  efficacy evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Junjie Wang, MD, Principal Investigator — Peking University 3rd Hospital radiation oncology department
Locations (1):
- Peking University 3rd Hospital, Beijing, Beijng, China

REFERENCES:
- [Derived] Jiang P, Wei S, Li C, Qu A, Chen H, Zhang H, Guo H, Wang J. Safety and efficacy of toripalimab plus concurrent chemoradiotherapy for locally advanced cervical cancer: a single-arm, phase Ib trial. BMC Cancer. 2025 Oct 14;25(1):1566. doi: 10.1186/s12885-025-15059-y. PMID 41087995